CLINICAL TRIAL: NCT03698695
Title: A Double Blind, Placebo-controlled, Randomized, 15-day Treatment, Pharmacodynamics, Safety, and Pharmacokinetics Study of THN201 Versus Donepezil Administered Orally to Healthy Male Volunteers Including a Scopolamine Challenge
Brief Title: A Pharmacodynamics, Safety, and Pharmacokinetics Study of THN201 Versus Donepezil in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theranexus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: THN201-101
Record Dates: First submitted 2018-10-02; First posted 2018-10-09 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Donepezil; Mefloquine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- THN201 (Experimental): THN201: Donepezil 5mg capsule and Mefloquine 10mg capsule once daily for 15 days
  Interventions: Drug: THN 201
- Donepezil (Active Comparator): Donepezil 5mg capsule and Mefloquine placebo capsule once daily for 15 days
  Interventions: Drug: Donepezil
- Placebo (Placebo Comparator): Donepezil placebo capsule and Mefloquine placebo capsule once daily for 15 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: THN 201 — THN 201: Donepezil 5 mg and Mefloquine 10 mg/d
  Other Names: Donepezil; Mefloquine
  Arms: THN201
Drug: Donepezil — Donepezil 5 mg/d and Mefloquine placebo
  Arms: Donepezil
Drug: Placebo — Donepezil placebo and Mefloquine placebo
  Arms: Placebo

SUMMARY:
This study explores the safety, pharmacodynamics and pharmacokinetics of THN201 a combination of donepezil and mefloquine to improve cognitive function in healthy male volunteers after impairment by a scopolamine challenge.

DETAILED DESCRIPTION:
This is a double-blind, 3-arm, parallel group study of 15 days duration including a scopolamine challenge at D15. Healthy male subjects will receive daily doses of THN201 (donepezil 5 mg and mefloquine), donepezil 5 mg or placebo and one subcutaneous injection of scopolamine 0.5 mg on D15. Cognitive function, EEG and P300 will be assessed at baseline and before and after scopolamine challenge at D15. A final safety evaluation will be performed 2 weeks after the end of the treatment period. Pharmacokinetic assessments will be performed to obtain a time/concentration profile of donepezil and mefloquine.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (BMI), calculated as weight in kg/(height in m)², from 18 to 30 kg/m², inclusive
* Healthy as determined by the investigator after a comprehensive clinical assessment based on medical history, physical examination, clinical laboratory test results, vital sign measurements, blood pressure (BP), heart rate (HR) and digital 12-lead ECG readings (all results should be normal or, if out of range, they should be non-clinically significant as determined by the investigator)

Exclusion Criteria:

* Any significant cardiovascular (e.g. heart failure), pulmonary (including asthma), hepatic, renal, respiratory (e.g. asthma), gastrointestinal, endocrine (e.g. diabetes, dyslipidaemia), immunologic, dermatological, haematological, neurologic, psychiatric disease, history of any clinically important drug allergy, systemic or presence of infectious disease.
* Current suicide risk or history of suicide risk (C-SSRS baseline: "yes" answer to items 4 and/or 5).
* Brain imaging (MRI) at screening showing anatomical or vascular abnormality of any type.
* EEG examination at screening showing abnormal (epileptiform) activities.
* Symptomatic hypotension,
* Participants with, or with a history of cardiac arrhythmia or cardiac disease or a personal or family history of long QT syndrome or a family history of sudden death.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* Antimalarial medicine intake or returning from a malaria-endemic area within the 12 last months before the first IMP administration.
* Planning to visit a country requiring antimalarial chemoprophylaxis during the study period.
* History of adverse reaction after a previous mefloquine intake.
* Contraindication for the use of Aricept® or for one of its excipients.
* Contraindication for the use of piperidine derivative compounds or for other cholinesterase inhibitors.
* Contraindication for the use of Lariam® or for one of its excipients.
* Contraindication for the use of scopolamine S.C. injection.
* History or presence of drug or alcohol abuse (alcohol consumption > 21 units / week).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics: Cognitive function measured with the Cognitive Drug Research (CDR) test battery | 15 days
  Main variable: Power of attention is the sum of the speed scores (msec) from three tests: Simple Reaction Time, Choice Reaction Time, and Digital Vigilance. Low values indicate better performance

SECONDARY OUTCOMES:
Safety Adverse events | 29 days
  Number of subjects with spontaneously reported treatment related adverse events

OTHER OUTCOMES:
Pharmacokinetics Plasma concentration of donepezil and mefloquine | 29 days
  Time profile of plasma concentrations of donepezil and mefloquine
Pharmacodynamics measured by quantitative EEG (qEEG) | 15 days
  Spectral analysis of absolute and/or relative amplitude in delta, theta, alpha, beta and gamma bands;
Pharmacodynamics measured by event related EEG potentials (P300) | 15 days
  Auditory P300 parameters (amplitude, latency and AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Régis Bordet, Prof., Principal Investigator — CHU Lille
Locations (7):
- France (7):
  - CHU Bordeaux, Bordeaux
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - CHU Lille, Lille
  - CHU Marseille, Marseille
  - Biotrial, Rennes
  - CHU Toulouse, Toulouse